CLINICAL TRIAL: NCT05514431
Title: Conversion of Labor Analgesia for Intrapartum Cesarean Delivery: Dural Puncture Epidural vs Combined Spinal Epidural vs Epidural
Brief Title: Conversion of Labor Analgesia for Intrapartum Cesarean Delivery: DPE v CSE v Epidural
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Emily E. Sharpe, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 20-004677
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia; Analgesia
Keywords: epidural; cesarean; parturient
MeSH Terms: conditions — Agnosia | interventions — Injections, Epidural; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Dural puncture epidural (DPE): Subjects that received neuraxial labor analgesia of dural puncture epidural for intrapartum cesarean delivery
  Interventions: Procedure: Dural Puncture Epidural (DPE) technique
- Combined spinal epidural (CSE): Subjects that received neuraxial labor analgesia of combined spinal epidural for intrapartum cesarean delivery
  Interventions: Procedure: Combined Spinal-Epidural (CSE) technique
- Traditional Epidural: Subjects that received neuraxial labor analgesia of epidural for intrapartum cesarean delivery
  Interventions: Procedure: Epidural

INTERVENTIONS:
Procedure: Epidural — Traditional epidural catheter placement
  Groups: Traditional Epidural
Procedure: Dural Puncture Epidural (DPE) technique — Epidural catheters placed via DPE technique
  Groups: Dural puncture epidural (DPE)
Procedure: Combined Spinal-Epidural (CSE) technique — Epidural catheters placed via CSE technique
  Groups: Combined spinal epidural (CSE)

SUMMARY:
As the dural puncture epidural (DPE) is increasing in popularity for labor analgesia, it is important to understand how it impacts outcomes in parturients. Prior studies have found epidural catheters placed via the combined-spinal epidural technique have greater success at surgical conversion for cesarean delivery than catheters placed via traditional techniques. The investigators aim to determine if epidural catheters placed by a DPE technique will also have an increased successful conversion for surgical anesthesia by conducting a retrospective review of all CD during the study period. If an association is found, this could be another benefit of DPE for labor analgesia.

DETAILED DESCRIPTION:
Electronic medical records will be searched for all intrapartum cesarean deliveries performed from February 1, 2017 through May 30, 2021 (Mayo Clinic) and from January 1, 2022 to December 31, 2022 (BC Women's Hospital).

From this list, patients that had cesarean delivery with an epidural catheter will be identified and split into three groups based on the type of neuraxial block listed in the block document of the patient's medical record:

Group 1 - Dural puncture epidural Group 2 - Epidural Group 3 - Combined spinal-epidural

Failure of epidural catheter conversion to surgical anesthesia at cesarean delivery will be defined by requirement of a second anesthetic at the time of surgery, including spinal or repeat epidural techniques or general anesthesia at the time of cesarean delivery

Data Collection: All data will be collected retrospectively from the electronic medical record.

1. Type of neuraxial block
2. Size of needle used for DPE or CSE: 25 g or 27 g
3. Duration of time from epidural placement until CD (Time of epidural placement; time of delivery)
4. Number of epidural top-ups
5. Type and amount of medication used for conversion to surgical anesthesia
6. Urgency of cesarean delivery
7. Airway documentation indicative of general anesthesia (if applicable)
8. Length (time) of surgical procedure

Other data collected from patient electronic records will include:

1. Maternal demographics: Parity, number of prior cesarean deliveries, weight, height, BMI
2. Fetal characteristics (birthweight, Apgar scores)
3. Indication for cesarean delivery

   1. Fetal distress (NRFHT, fetal intolerance of labor)
   2. Failure of labor (Failure to dilate, failure to descend)
   3. Failed operative vaginal delivery
   4. Maternal comorbidity
   5. Emergency (cord prolapse, abruption, uterine rupture)
4. Anesthesiologist (Fellowship trained: Y/N) at time of cesarean delivery

ELIGIBILITY:
Inclusion Criteria:

1. Women with neuraxial labor analgesia (CSE, DPE, or Epidural) who have an intrapartum cesarean delivery
2. Singleton gestation

Exclusion Criteria:

1. No local anesthetic given in epidural for cesarean delivery (in emergency situation)
2. Inadvertent dural puncture

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parturients that undergo intrapartum cesarean delivery with an epidural already in situ.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Conversion to surgical anesthesia | Baseline
  Number of subject to have success of conversion to surgical anesthesia for intrapartum cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Emily Sharpe, MD, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials